CLINICAL TRIAL: NCT01292226
Title: Relationships Between Pharmacokinetic and Pharmacodynamic Strategies for Assessment of the Risks for Acute Rejection and Side Effects of Mycophenolate Mofetil
Brief Title: A Study of the Correlation Between Pharmacokinetic and Pharmacodynamic Parameters of CellCept (Mycophenolate Mofetil).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML19835
Record Dates: First submitted 2011-02-03; First posted 2011-02-09 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-04

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Mycophenolic Acid; Cyclosporine; Adrenal Cortex Hormones

ARMS (1):
- Mycophenolate Mofetil Monotherapy (Experimental): Participants received an initial dose of mycophenolate mofetil (MMF), 1 gram (g), orally (PO), twice per day (BID), within 5 days of transplant for 24 weeks. Participants also received concurrent antibody induction, cyclosporine, and corticosteroids as needed according to center's practice.
  Interventions: Drug: mycophenolate mofetil; Drug: antibody induction; Drug: Cyclosporine; Drug: corticosteroid

INTERVENTIONS:
Drug: mycophenolate mofetil — 1 g PO BID for 24 weeks
  Other Names: CellCept
Drug: antibody induction — According to manufacturer recommendation
Drug: Cyclosporine — According to manufacturer recommendation
Drug: corticosteroid — According to manufacturer recommendation

SUMMARY:
This study will evaluate the correlation between the pharmacokinetic and pharmacodynamic parameters of CellCept in patients undergoing primary kidney transplantation, in order to assess the impact on clinical outcome and the risks of acute rejection. All patients will receive oral CellCept, 1g twice daily, and pharmacokinetic and pharmacodynamic parameters will be measured at weeks 2, 4, 12 and 24. The anticipated time on study treatment is 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 to 65 years of age
* Patients undergoing primary kidney transplantation

Exclusion Criteria:

* Recipients of multiple organ transplants
* Prior therapy with CellCept
* Presence or history of malignancies, except for successfully treated basal or squamous cell carcinoma of the skin
* Active peptic ulcer or active serious digestive system disease that may affect the absorption of CellCept

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (7):
- Italy (7):
  - Bari
  - Brescia
  - Coppito
  - Napoli
  - Roma
  - Torino
  - Verona

RESULTS

PARTICIPANT FLOW:
Groups:
- Mycophenolate Mofetil (MMF) Monotherapy: Participants received an initial dose of MMF 1 gram (g), orally (PO), twice per day (BID), started within 5 days of transplant, for up to 24 weeks. MMF dose could be titrated to a maximum daily dose of 2 g (minimum daily dose was 1 g). Participants also received concurrent antibody induction, cyclosporine, and corticosteroids as needed according to center's practice.
Period: Overall Study
Arm/Group | Mycophenolate Mofetil (MMF) Monotherapy
Started | 45
Completed | 32
Not Completed | 13
Not completed — Adverse Event | 5
Not completed — Death | 1
Not completed — Graft loss | 1
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- MMF Monotherapy: Participants received an initial dose of MMF 1 g, PO, BID, started within 5 days of transplant, for up to 24 weeks. MMF dose could be titrated to a maximum daily dose of 2 g (minimum daily dose was 1 g). Participants also received concurrent antibody induction, cyclosporine, and corticosteroids as needed according to center's practice.
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.60 (9.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Acute Rejection
Description: Diagnosis of acute rejection was suspected in any participant with an increase in serum creatinine greater than or equal to (≥) 25 percent (%). All suspected acute rejections were confirmed by biopsy. The start date of acute rejection was identified as the date of biopsy.
Time Frame: Day 1, Weeks 2, 4, 12, 24, and 28
Population: Intent-to-treat (ITT) population: all eligible participants who had at least baseline (BL) and 1 assessment of pharmacokinetics (PK) and pharmacodynamics (PD). Acute rejection was analyzed in any participant with an increase in serum creatinine of 25%.
Measure: Number; unit: percentage of participants
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
percentage of participants | 9.1

2. Primary Outcome: Time to Rejection
Description: The mean time, in days, from the date of enrollment to date of biopsy confirming acute rejection.
Time Frame: Day 1, Weeks 2, 4, 12, 24, and 28
Population: ITT population; only participants with acute or biopsy-proven rejection were included in the analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 6
days | 23.67 (21.44)

3. Secondary Outcome: Percentage of Participants With Graft Loss
Description: An allograft was presumed to be lost if a participant started dialysis and was not able to subsequently be removed from dialysis.
Time Frame: Day 1, Weeks 2, 4, 12, 24, and 28
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
percentage of participants | 2.3

4. Secondary Outcome: Percentage of Participants Surviving
Time Frame: Day 1, Weeks 2, 4, 12, 24, and 28
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
percentage of participants | 97.7

5. Secondary Outcome: Total Mycophenolate Acid (MPA) by Visit and Timepoint
Description: Drug quantification of total MPA (micrograms per milliliter [mcg/mL]) in the plasma was measured at time (T) = 0 minutes (min), 40 mins, and 120 mins.
Time Frame: Weeks 2, 4, 12, 24, and 28 (Safety Follow-Up Visit), and any unscheduled visits
Population: ITT population; n=number of samples analyzed.
Measure: Mean (Standard Deviation); unit: mcg/mL
Units Other Than Participants: Samples
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
Number analyzed (Samples) | 491
mcg/mL
  T=0, Week 2 (n=41) | 1.75 (1.49)
  T=0, Week 4 (n=42) | 1.87 (1.62)
  T=0, Week 12 (n=35) | 1.79 (1.04)
  T=0, Week 24 (n=35) | 1.90 (1.53)
  T=0, safety follow-up (n=3) | 1.16 (0.22)
  T=0, unscheduled visit (n=7) | 1.32 (0.67)
  T=0, overall mean value (n=163) | 1.79 (1.40)
  T=40, Week 2 (n=43) | 6.44 (4.37)
  T=40, Week 4 (n=42) | 6.96 (3.92)
  T=40, Week 12 (n=35) | 7.23 (4.27)
  T=40, Week 24 (n=35) | 6.47 (3.35)
  T=40, safety follow-up (n=3) | 5.71 (0.55)
  T=40, unscheduled visit (n=7) | 4.06 (1.05)
  T=40, overall mean value (n=165) | 6.63 (3.91)
  T=120, Week 2 (n=41) | 8.86 (7.30)
  T=120, Week 4 (n=42) | 8.95 (6.33)
  T=120, Week 12 (n=35) | 8.57 (6.71)
  T=120, safety follow-up (n=3) | 4.91 (2.09)
  T=120, Week 24 (n=35) | 10.04 (6.91)
  T=120, unscheduled visit (n=7) | 7.03 (5.31)
  T=120, overall mean value (n=163) | 8.92 (6.68)

6. Secondary Outcome: Free MPA (mcg/mL) by Visit
Description: Drug quantification of free MPA in the plasma was measured at T = 0, 40, and 120 mins.
Time Frame: Weeks 2, 4, 12, 24, safety follow-up (Week 28), and any unscheduled visits
Population: ITT population; n=number of samples analyzed.
Measure: Mean (Standard Deviation); unit: mcg/mL
Units Other Than Participants: Samples
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
Number analyzed (Samples) | 482
mcg/mL
  T=0, Week 2 (n=40) | 0.03 (0.03)
  T=0, Week 4 (n=39) | 0.04 (0.03)
  T=0, Week 12 (n=33) | 0.03 (0.02)
  T=0, Week 24 (n=32) | 0.03 (0.02)
  T=0, safety follow-up (n=3) | 0.01 (0.01)
  T=0, unscheduled visit (n=7) | 0.04 (0.03)
  T=0, overall mean value (n=154) | 0.03 (0.03)
  T=40, Week 2 (n=41) | 0.11 (0.09)
  T=40, Week 4 (n=42) | 0.11 (0.07)
  T=40, Week 12 (n=35) | 0.11 (0.06)
  T=40, Week 24 (n=35) | 0.38 (1.35)
  T=40, safety follow-up (n=3) | 0.06 (0.02)
  T=40, unscheduled visit (n=7) | 0.09 (0.07)
  T=40, overall mean value (n=163) | 0.17 (0.63)
  T=120, Week 2 (n=43) | 0.11 (0.07)
  T=120, Week 4 (n=42) | 0.11 (0.07)
  T=120, Week 12 (n=35) | 0.16 (0.36)
  T=120, Week 24 (n=35) | 0.10 (0.06)
  T=120, safety follow-up (n=3) | 0.10 (0.03)
  T=120, unscheduled visit (n=7) | 0.07 (0.03)
  T=120, overall mean value (n=165) | 0.12 (0.18)

7. Primary Outcome: Percentage of Participants With Biopsy-Proven Acute Rejection (BPAR)
Description: BPAR was defined according to 1997 Banff Criteria as a biopsy Banff grade of IA, IB, IIA, IIB, or III. Grade IA was defined as significant interstitial infiltration with greater than (>)25% of parenchyma affected, and foci of moderate tubulitis with >4 mononuclear cells per tubular cross section or group of 10 tubular cells. Grade IB was defined as significant interstitial infiltration with >25% parenchyma affected, and foci of severe tubulitis with >10% mononuclear cells per tubular cross section or group of 10 tubular cells. Grade IIA was defined as mild to moderate intimal arteritis. Grade IIB was defined as severe intimal arteritis comprising >25% of the luminal area. Grade III was defined as transmural arteritis and/or arterial fibrinoid changes and necrosis of medial smooth muscle cells.
Time Frame: Day 1, Weeks 2, 4, 12, 24, and 28
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
percentage of participants | 4.5

8. Secondary Outcome: MPA Area Under the Concentration - Time Curve From Time 0 to 12 Hours (AUC0-12) (mcg/mL) by Visit
Description: The AUC0-12 of MPA was estimated on the validated limited sampling strategy, AUC (milligrams multiplied by height over liter [mg.h/L]) = 7.182 + 4.607 multiplied by (*) concentration at 0 minutes (C0)+ 0.998 * the concentration at 40 minutes (C0.67) + 2.149 * the concentration at 120 minutes (C2).
Time Frame: Predose and 40 minutes and 2 hours postdose at Weeks 2, 4, 12, and 24, and at the Safety follow-up (Week 28)
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
mcg*hr/mL
  Week 2 (n=41) | 38.3 (17.9)
  Week 4 (n=42) | 39.7 (17.4)
  Week 12 (n=35) | 39.7 (16.5)
  Week 24 (n=35) | 39.8 (17.0)
  Follow-up (n=3) | 29.7 (3.7)

9. Secondary Outcome: Inosine MonoPhosphate DeHydrogenase (IMPDH) Activity by Visit and Timepoint
Description: IMPDH activity in peripheral blood mononuclear cells (PBMCs) was measured at 2 timepoints per visit, 0 and 120 minutes and presented in enzyme units. The unit of measure of enzyme activity is "U". One U is defined as the amount of the enzyme that produces a certain amount of enzymatic activity that is, the amount that catalyzes the conversion of 1 micro mole of substrate per minute under pre-specified conditions (temperature, pH).
Time Frame: BL and Weeks 2, 4, 12, and 24, and safety follow-up (Week 28) and any unscheduled visits
Population: ITT population; n=number of samples analyzed.
Measure: Mean (Standard Deviation); unit: enzyme units
Units Other Than Participants: Samples
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
Number analyzed (Samples) | 364
enzyme units
  T=0, BL (n=44) | 5.01 (5.17)
  T=0, Week 2 (n=42) | 3.96 (3.58)
  T=0, Week 4 (n=42) | 3.89 (2.36)
  T=0, Week 12 (n=35) | 6.74 (11.79)
  T=0, Week 24 (n=34) | 9.58 (10.81)
  T=0, safety follow-up (n=0) | 0 (0)
  T=0, unscheduled visit (n=7) | 6.00 (6.12)
  T=0, mean value (n=204) | 5.65 (7.54)
  T=120, BL (n=0) | 0 (0)
  T=120, Week 2 (n=42) | 3.06 (3.42)
  T=120, Week 4 (n=42) | 3.10 (2.66)
  T=120, Week 12 (n=35) | 3.75 (5.02)
  T=120, Week 24 (n=34) | 6.39 (6.14)
  T=120, safety follow-up (n=0) | 0 (0)
  T=120, unscheduled visit (n=7) | 3.89 (1.82)
  T=120, mean value (n=160) | 3.97 (4.46)

10. Secondary Outcome: IMPDH Expression I by Visit and Timepoint
Description: IMPDH I gene expression was measured by real time polymerase chain reaction (QRT-PCR) based cytokine measurement of PBMCs at 2 timepoints per visit, 0 and 120 minutes and expressed as number of messenger ribonucleic acid (mRNA) copies per cell (copies/cell).
Time Frame: BL and Weeks 2, 4, 12, and 24, and safety follow-up (Week 28) and any unscheduled visits
Population: ITT population; n=number of samples analyzed.
Measure: Mean (Standard Deviation); unit: number of mRNA copies/cell
Units Other Than Participants: Samples
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
Number analyzed (Samples) | 369
number of mRNA copies/cell
  T=0, BL (n=44) | 2.32 (3.02)
  T=0, Week 2 (n=41) | 32.29 (188.29)
  T=0, Week 4 (n=42) | 3.16 (8.59)
  T=0, Week 12 (n=34) | 4.10 (15.09)
  T=0, Week 24 (n=34) | 1.95 (2.94)
  T=0, safety follow-up (n=3) | 11803.48 (20432.48)
  T=0, unscheduled visit (n=7) | 4.00 (3.84)
  T=0, mean value (n=205) | 181.48 (2473.05)
  T=120, BL (n=0) | 0 (0)
  T=120, Week 2 (n=43) | 4146.17 (14891.57)
  T=120, Week 4 (n=42) | 1692.11 (6690.21)
  T=120, Week 12 (n=35) | 1556.06 (5856.17)
  T=120, Week 24 (n=34) | 3.02 (7.53)
  T=120, safety follow-up (n=3) | 107.30 (179.38)
  T=120, unscheduled visit (n=7) | 1038.52 (1781.89)
  T=120, mean value (n=164) | 1899.45 (8824.89)

11. Secondary Outcome: IMPDH Expression II by Visit and Timepoint
Description: IMPDH II gene expression was measured by QRT-PCR based cytokine measurement of PBMCs at 2 timepoints per visit, 0 and 120 minutes and expressed as number of mRNA copies/cell.
Time Frame: BL and Weeks 2, 4, 12, and 24, and safety follow-up (Week 28) and any unscheduled visits
Population: ITT population; n=number of samples analyzed.
Measure: Mean (Standard Deviation); unit: number of mRNA copies/cell
Units Other Than Participants: Samples
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
Number analyzed (Samples) | 369
number of mRNA copies/cell
  T=0, BL (n=44) | 115.33 (19.81)
  T=0, Week 2 (n=41) | 113.43 (21.67)
  T=0, Week 4 (n=42) | 117.16 (30.72)
  T=0, Week 12 (n=34) | 112.43 (24.57)
  T=0, Week 24 (n=34) | 114.21 (19.79)
  T=0, safety follow-up (n=3) | 123.86 (37.61)
  T=0, unscheduled visit (n=7) | 116.57 (19.25)
  T=0, mean value (n=205) | 114.82 (23.54)
  T=120, BL (n=0) | 0 (0)
  T=120, Week 2 (n=43) | 304.64 (309.26)
  T=120, Week 4 (n=42) | 148.32 (206.39)
  T=120, Week 12 (n=35) | 143.11 (82.95)
  T=120, Week 24 (n=34) | 109.00 (22.81)
  T=120, safety follow-up (n=3) | 140.51 (42.37)
  T=120, unscheduled visit (n=7) | 167.19 (155.73)
  T=120, mean value (n=164) | 180.71 (208.68)

12. Secondary Outcome: Interleukin 8 (IL-8) Expression by Visit and Timepoint
Description: IL-8 gene expression was measured by QRT-PCR based cytokine measurement of PBMCs at 2 timepoints per visit, 0 and 120 minutes and expressed as number of mRNA copies/cell.
Time Frame: BL and Weeks 2, 4, 12, and 24, and safety follow-up (Week 28) and any unscheduled visits
Population: ITT population; n=number of samples analyzed.
Measure: Mean (Standard Deviation); unit: number of mRNA copies/cell
Units Other Than Participants: Samples
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
Number analyzed (Samples) | 369
number of mRNA copies/cell
  T=0, BL (n=44) | 4532.72 (11598.93)
  T=0, Week 2 (n=41) | 29960.41 (128979.24)
  T=0, Week 4 (n=42) | 54101.30 (262581.32)
  T=0, Week 12 (n=34) | 1829.87 (6411.17)
  T=0, Week 24 (n=34) | 10391.60 (42574.52)
  T=0, safety follow-up (n=3) | 1254.29 (1150.40)
  T=0, unscheduled visit (n=7) | 19148.94 (49991.25)
  T=0, mean value (n=205) | 20748.32 (1333817.10)
  T=120, BL (n=0) | 0.0 (0.0)
  T=120, Week 2 (n=43) | 1028.93 (4210.43)
  T=120, Week 4 (n=42) | 21227.11 (103517.73)
  T=120, Week 12 (n=35) | 12022.83 (63647.48)
  T=120, Week 24 (n=34) | 9418.65 (29084.00)
  T=120, safety follow-up (n=3) | 397887.30 (688477.81)
  T=120, unscheduled visit (n=7) | 220.14 (457.26)
  T=120, mean value (n=164) | 17512.31 (110920.39)

13. Secondary Outcome: Tumor Necrosis Factor (TNF) Expression by Visit and Timepoint
Description: TNF gene expression was measured by QRT-PCR based cytokine measurement of PBMCs at 2 timepoints per visit, 0 and 120 minutes and expressed as number of mRNA copies/cell.
Time Frame: BL and Weeks 2, 4, 12, and 24, and safety follow-up (Week 28) and any unscheduled visits
Population: ITT population; n=number of samples analyzed.
Measure: Mean (Standard Deviation); unit: number of mRNA copies/cell
Units Other Than Participants: Samples
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
Number analyzed (Samples) | 369
number of mRNA copies/cell
  T=0, BL (n=44) | 4532.72 (11598.93)
  T=0, Week 2 (n=41) | 29960.41 (128979.24)
  T=0, Week 4 (n=42) | 54101.30 (262581.32)
  T=0, Week 12 (n=34) | 1829.87 (6411.17)
  T=0, Week 24 (n=34) | 10391.60 (42574.52)
  T=0, safety follow-up (n=3) | 1254.29 (1150.40)
  T=0, unscheduled visit (n=7) | 19148.94 (49991.25)
  T=0, mean value (n=205) | 20748.32 (133817.10)
  T=120, BL (n=0) | 0 (0)
  T=120, Week 2 (n=43) | 1028.93 (4210.43)
  T=120, Week 4 (n=42) | 21227.11 (103517.73)
  T=120, Week 12 (n=35) | 12022.83 (63647.48)
  T=120, Week 24 (n=34) | 9418.65 (29084.00)
  T=120, safety follow-up (n=3) | 397887.30 (688477.81)
  T=120, unscheduled visit (n=7) | 220.14 (457.26)
  T=120, mean value (n=164) | 17512.31 (110920.39)

14. Secondary Outcome: Percentage of Participants With Infection
Description: Infections were graded according to the World Health Organization (WHO) worst grade observed.
Time Frame: BL and Weeks 2, 4, 12, 24, and 28 (Safety Follow-Up)
Population: Safety population: all enrolled participants
Measure: Number; unit: percentage of participants
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 45
percentage of participants
  Acarodermatitis (mild) | 2.22
  Bronchitis (moderate) | 2.22
  Cytomegalovirus (CMV) infection (mild) | 13.33
  CMV infection (moderate) | 8.89
  CMV infection (severe) | 4.44
  CMV viraemia (mild) | 2.22
  Gastroenteritis proteus (severe) | 2.22
  Gastrointestinal infection (severe) | 2.22
  Legionella infection (life-threatening) | 2.22
  Oral herpes (mild) | 2.22
  Sepsis (life-threatening) | 2.22
  Tracheitis (mild) | 2.22
  Urethritis (mild) | 2.22
  Urinary tract infection (mild) | 28.89
  Urinary tract infection (moderate) | 2.22

15. Secondary Outcome: Percentage of Participants With Gastrointestinal Toxicities
Description: Gastrointestinal adverse events (AEs) according to WHO worst grade observed.
Time Frame: BL and Weeks 2, 4, 12, 24, and 28 (Safety Follow-up Visit)
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 45
percentage of participants
  Abdominal pain (moderate) | 2.22
  Abdominal pain (severe) | 2.22
  Anal fissure (mild) | 2.22
  Diarrhoea (mild) | 4.44
  Diarrhoea (moderate) | 2.22
  Diarrhoea (severe) | 2.22
  Dyspepsia (mild) | 2.22
  Gastritis (moderate) | 2.22
  Gastritis erosive (moderate) | 2.22
  Gingival hyperplasia (mild) | 2.22
  Haemorrhoids (mild) | 2.22
  Intra-abdominal haematoma (mild) | 2.22
  Nausea (moderate) | 2.22
  Stomatitis (mild) | 2.22
  Vomiting (mild) | 2.22
  Vomiting (moderate) | 4.44
  Vomiting (severe) | 4.44

16. Secondary Outcome: Percentage of Participants With Hematologic Toxicity
Description: Hematological toxicities graded according to WHO worst grade observed (Grade 1=mild, Grade 2=moderate).
Time Frame: BL and Weeks 2, 4, 12, 24, and 28 (Safety Follow-Up)
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 45
percentage of participants
  Grade 1 hemoglobin decreased | 13.33
  Grade 1 leukocytes decreased | 11.11
  Grade 2 leukocytes decreased | 8.89
  Grade 1 granulocytes decreased | 6.67
  Grade 2 granulocytes decreased | 6.67
  Grade 1 platelets decreased | 6.67
  Grade 1 bilirubin increased | 4.44
  Grade 2 bilirubin increased | 2.22
  Grade 1 hypoglycemia | 4.44
  Grade 1 alkaline phosphatase increased | 13.33
  Grade 2 alkaline phosphatase increased | 2.22
  Grade 1 aspartate aminotransferase increased | 6.67
  Grade 1 alanine aminotransferase increased | 8.89
  Grade 2 alanine aminotransferase increased | 2.22
  Grade 1 cholesterol increased | 26.67
  Grade 2 cholesterol increased | 8.89
  Grade 1 triglycerides increased | 24.44
  Grade 2 triglycerides increased | 2.22
  Grade 1 blood urea nitrogen increased | 2.22
  Grade 2 blood urea nitrogen increased | 2.22

17. Secondary Outcome: Spearman's Rank Correlation Coefficient Between MPA Levels and IMPDH Activity
Description: The Spearman's rank correlation coefficient was computed by ranking the data from 2 time points, 0 minutes and 120 minutes, and using the ranks in the Pearson product-moment correlation formula. In case of ties, the averaged ranks were used.
Time Frame: BL and Weeks 2, 4, 12, and 24
Population: ITT population; n=number of samples analyzed.
Measure: Number; unit: correlation coefficient
Units Other Than Participants: Samples
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
Number analyzed (Samples) | 305
correlation coefficient
  Free MPA, T=0 (n=144) | 0.063
  Free MPA, T=120 (n=153) | 0.028
  Total MPA, T=0 (n=152) | 0.034
  Total MPA, T=120 (n=153) | -0.050
Statistical Analysis 1: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.4505, ANOVA — Free MPA, time 0 [trough]; Analysis of variance (ANOVA)
Statistical Analysis 2: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.7322, ANOVA — Free MPA, time 120 [2 hours after administration at Week 12]
Statistical Analysis 3: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.6798, ANOVA — Total MPA, time 0 [trough]
Statistical Analysis 4: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.5410, ANOVA — Total MPA, time 120 [2 hours after administration at Week 12]

18. Secondary Outcome: Spearman's Rank Correlation Coefficient Between IMPDH I Expression and MPA Levels
Description: as for outcome 17
Time Frame: BL and Weeks 2, 4, 12, and 24
Population: ITT population; n=number of samples analyzed
Measure: Number; unit: correlation coefficient
Units Other Than Participants: Samples
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
Number analyzed (Samples) | 290
correlation coefficient
  Free MPA, T=0 (n=141) | 0.073
  Free MPA, T=120 (n=143) | -0.024
  Total MPA, T=0 (n=147) | 0.037
  Total MPA, T=120 (n=143) | -0.140
Statistical Analysis 1: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.3892, ANOVA — Free MPA, time 0 [trough]
Statistical Analysis 2: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.6564, ANOVA — Total MPA, time 0 [trough]
Statistical Analysis 3: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.7772, ANOVA — Free MPA, time 120 [2 hours after administration at Week 12]
Statistical Analysis 4: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.0958, ANOVA — Total MPA, time 120 [2 hours after administration at Week 12]

19. Secondary Outcome: Spearman's Rank Correlation Coefficient Between IMPDH I Expression and Free Fraction
Description: as for outcome 17
Time Frame: BL and Weeks 2, 4, 12, and 24
Population: ITT population; n=number of samples analyzed.
Measure: Number; unit: correlation coefficient
Units Other Than Participants: Samples
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
Number analyzed (Samples) | 283
correlation coefficient
  p Free fraction, T=0 (n=140) | 0.047
  p Free fraction, T=120 (n=143) | 0.080
Statistical Analysis 1: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.5796, ANOVA — Time 0 [trough]
Statistical Analysis 2: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.3428, ANOVA — Time 120 [2 hours after administration at Week 12]

20. Secondary Outcome: Spearman's Rank Correlation Coefficient Between IMPDH II Expression and MPA Levels
Description: as for outcome 17
Time Frame: BL and Weeks 2, 4, 12, and 24
Population: ITT population; n=number of samples analyzed.
Measure: Number; unit: correlation coefficient
Units Other Than Participants: Samples
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
Number analyzed (Samples) | 305
correlation coefficient
  Free MPA, T=0 (n=145) | 0.007
  Free MPA, T=120 (n=153) | 0.073
  Total MPA, T=0 (n=152) | -0.001
  Total MPA, T=120 (n=153) | 0.084
Statistical Analysis 1: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.9372, ANOVA — Free MPA, time 0 [trough]
Statistical Analysis 2: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.9904, ANOVA — Total MPA, time 0 [trough]
Statistical Analysis 3: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.3658, ANOVA — Free MPA, time 120 [2 hours after administration at Week 12]
Statistical Analysis 4: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.2987, ANOVA — Total MPA, time 120 [2 hours after administration at Week 12]

21. Secondary Outcome: Spearman's Rank Correlation Coefficient Between IMPDH II Expression and Free Fraction
Description: as for outcome 17
Time Frame: BL and Weeks 2, 4, 12, and 24
Population: ITT population; n=number of samples analyzed.
Measure: Number; unit: correlation coefficient
Units Other Than Participants: Samples
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
Number analyzed (Samples) | 297
correlation coefficient
  p Free fraction, T=0 (n=144) | -0.027
  p Free fraction, T=120 (n=153) | 0.015
Statistical Analysis 1: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.7455, ANOVA — time 0 [trough]
Statistical Analysis 2: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.8504, ANOVA — Time 120 [2 hours after administration at Week 12]

22. Secondary Outcome: Spearman's Rank Correlation Coefficient Between IMPDH Inhibition and Risk of Acute Rejection
Description: as for outcome 17
Time Frame: BL and Weeks 2, 4, 12, and 24
Population: ITT population; n=number of samples analyzed.
Measure: Number; unit: correlation coefficient
Units Other Than Participants: Samples
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
Number analyzed (Samples) | 353
correlation coefficient
  IMPDH I expression, T=0 (n=189) | 0.030
  IMPDH I expression T=120 (n=145) | 0.083
  IMPDH II expression, T=0 (n=196) | -0.062
  IMPDH II expression (T=120, n=155) | -0.010
  MPDH Activity, T=0 (n=198) | -0.121
  IMPDH Activity, T=120 (n=155) | -0.004
Statistical Analysis 1: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.6847, ANOVA — IMPDH I, time 0 [trough]
Statistical Analysis 2: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.3184, ANOVA — IMPDH I, time 120 [2 hours after administration at Week 12]
Statistical Analysis 3: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.3862, ANOVA — IMPDH II, time 0 [trough]
Statistical Analysis 4: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.9040, ANOVA — IMPDH II, time 120 [2 hours after administration at Week 12]
Statistical Analysis 5: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.0907, ANOVA — IMPDH activity, time 0 [trough]
Statistical Analysis 6: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.9630, ANOVA — IMPDH activity, time 120 [2 hours after administration at Week 12]

23. Secondary Outcome: Spearman's Rank Correlation Coefficient Between IMPDH Expression and Risk of Infection
Description: as for outcome 17
Time Frame: BL and Weeks 2, 4, 12, and 24
Population: ITT population; n=number of samples analyzed.
Measure: Number; unit: correlation coefficient
Units Other Than Participants: Samples
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
Number analyzed (Samples) | 351
correlation coefficient
  IMPDH I expression (n=334) | 0.045
  IMPDH II expression (n=351) | 0.047
Statistical Analysis 1: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.4130, ANOVA — IMPDH I
Statistical Analysis 2: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.3823, ANOVA — IMPDH II

24. Secondary Outcome: Spearman's Rank Correlation Coefficient Between IMPDH Expression and Risk of Hematologic Toxicity
Description: as for outcome 17
Time Frame: BL and Weeks 2, 4, 12, and 24
Population: ITT population
Measure: Number; unit: correlation coefficient
Units Other Than Participants: Samples
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
Number analyzed (Samples) | 351
correlation coefficient
  IMPDH I expression (n=334) | -0.116
  IMPDH II expression (n=351) | -0.004
Statistical Analysis 1: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.0316, ANOVA — IMPDH I
Statistical Analysis 2: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.9440, ANOVA — IMPDH II

25. Secondary Outcome: Spearman's Rank Correlation Coefficient Between IMPDH Expression and Risk of Gastrointestinal Toxicity
Description: as for outcome 17
Time Frame: BL and Weeks 2, 4, 12, and 24
Population: ITT population
Measure: Number; unit: correlation coefficient
Units Other Than Participants: Samples
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
Number analyzed (Samples) | 351
correlation coefficient
  IMPDH I expression (n=334) | 0.082
  IMPDH II expression (n=351) | 0.030
Statistical Analysis 1: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.1328, ANOVA — IMPDH I
Statistical Analysis 2: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.5760, ANOVA — IMPDH II

26. Secondary Outcome: Spearman's Rank Correlation Coefficient Between MPA Levels and Risk of Infection
Description: as for outcome 17
Time Frame: BL and Weeks 2, 4, 12, and 24
Population: ITT population; n=number of samples
Measure: Number; unit: correlation coefficient
Units Other Than Participants: Samples
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
Number analyzed (Samples) | 308
correlation coefficient
  Free MPA (n=300) | -0.020
  Total MPA (n=308) | 0.063
  AUC MPA (n=152) | 0.030
Statistical Analysis 1: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.7332, ANOVA — Free MPA
Statistical Analysis 2: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.2681, ANOVA — Total MPA
Statistical Analysis 3: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.7087, ANOVA — AUC MPA

27. Secondary Outcome: Spearman's Rank Correlation Coefficient Between MPA Levels and Risk of Hematologic Toxicity
Description: as for outcome 17
Time Frame: BL and Weeks 2, 4, 12, and 24
Population: ITT population; n=number of samples
Measure: Number; unit: correlation coefficient
Units Other Than Participants: Samples
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
Number analyzed (Samples) | 308
correlation coefficient
  Free MPA (n=300) | -0.004
  Total MPA (n=308) | -0.037
  AUC MPA (n=152) | -0.038
Statistical Analysis 1: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.9432, ANOVA — Free MPA
Statistical Analysis 2: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.5177, ANOVA — Total MPA
Statistical Analysis 3: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.6398, ANOVA — AUC MPA

28. Secondary Outcome: Spearman's Rank Correlation Coefficient Between MPA Levels and Risk of Gastrointestinal Toxicity
Description: as for outcome 17
Time Frame: BL and Weeks 2, 4, 12, and 24
Population: ITT population; n=number of samples
Measure: Number; unit: correlation coefficient
Units Other Than Participants: Samples
Arm/Group | MMF Monotherapy
Number analyzed (Participants) | 44
Number analyzed (Samples) | 308
correlation coefficient
  Free MPA (n=300) | 0.106
  Total MPA (n=308) | 0.142
  AUC MPA (n=152) | 0.187
Statistical Analysis 1: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.0656, ANOVA — Free MPA
Statistical Analysis 2: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.0131, ANOVA — Total MPA
Statistical Analysis 3: Comparison: MMF Monotherapy; Test type: Superiority or Other; p = 0.0515, ANOVA — AUC MPA

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded throughout treatment to the safety evaluation follow up 4 weeks after treatment discontinuation, for up to 28 weeks.
Description: The safety assessment population included all eligible participants who received at least 1 dose of study treatment.
Arm/Group | MMF Monotherapy
Serious Adverse Events (participants affected / at risk) | 20/45
Other Adverse Events (participants affected / at risk) | 43/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MMF Monotherapy (N=45)
Acute renal failure (Renal and urinary disorders) | 1
CMV infection (Infections and infestations) | 3
Infection due to Legionella and Pseudomonas (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Tubulitis (Renal and urinary disorders) | 1
Ureteral stenosis (Renal and urinary disorders) | 1
Proteus mirabilis infection (Infections and infestations) | 1
Leucopenia (Blood and lymphatic system disorders) | 1
Urinary anastomotic leak (Renal and urinary disorders) | 1
Prostatic adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastrointestinal infection (Infections and infestations) | 1
Acute rejection (Injury, poisoning and procedural complications) | 3
Carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute vascular and interstitial rejection (Injury, poisoning and procedural complications) | 1
Lymphocele (Blood and lymphatic system disorders) | 15
Edema of the left leg (General disorders) | 1
Increase in creatinine (Investigations) | 2
Acute tubular necrosis (Renal and urinary disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MMF Monotherapy (N=45)
Urinary tract infection (Infections and infestations) | 22
Cytomegalovirus infection (Infections and infestations) | 9
Blood creatinine increased (Investigations) | 8
Blood cholesterol increased (Investigations) | 3
White blood cell count decreased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Vomiting (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Gastritis erosive (Gastrointestinal disorders) | 1
Gingival hyperplasia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 8
Hyperuricaemia (Metabolism and nutrition disorders) | 7
Hypercholesterolemia (Metabolism and nutrition disorders) | 4
Hyperlipemia (Metabolism and nutrition disorders) | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 1
Pyrexia (General disorders) | 12
Oedema peripheral (General disorders) | 4
Asthenia (General disorders) | 1
Catheter related infection (Infections and infestations) | 1
Hearing impaired (General disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 13
Anaemia (Blood and lymphatic system disorders) | 10
Lymphocele (Blood and lymphatic system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Antithrombin III deficiency (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Lymphocytopenia (Blood and lymphatic system disorders) | 1
Hypertension (Vascular disorders) | 6
Insomnia (Psychiatric disorders) | 5
Anxiety (Psychiatric disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Cholestasis (Hepatobiliary disorders) | 1
Erythema (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Renal colic (Renal and urinary disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Acarodermatitis (Skin and subcutaneous tissue disorders) | 1
Acidosis (Blood and lymphatic system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Lipidosis (Hepatobiliary disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Tracheitis (Infections and infestations) | 1
Urethritis (Infections and infestations) | 1
Wound haemorrhage (Surgical and medical procedures) | 1
Anal fissure (Gastrointestinal disorders) | 1
Arteriovenous fistula (Vascular disorders) | 1
Arteriovenous fistula thrombosis (Vascular disorders) | 1
Ear pain (General disorders) | 1
Coagulopathy (Blood and lymphatic system disorders) | 1
Cytomegalovirus viraemia (Infections and infestations) | 1
Glomerulosclerosis (Renal and urinary disorders) | 1
Operative haemorrhage (Surgical and medical procedures) | 1
Post-procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Intra-abdominal haematoma (Gastrointestinal disorders) | 1
Oral herpes (Gastrointestinal disorders) | 1
Pharyngolaryngeal pain (General disorders) | 1
Renal artery stenosis (Renal and urinary disorders) | 1
Perirenal haematoma (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.